CLINICAL TRIAL: NCT07059520
Title: Translesional PRESSURE Measurements to Assess Clinical Relevance of a Mesenteric Artery Stenosis (PRESSURE-study)
Acronym: PRESSURE
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Kay Pieterman, Radiologist, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC-2024-0491 / 12330
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chronic Mesenteric Ischemia; Ischemia, Mesenteric
Keywords: chronic mesenteric ischemia; Pd/Pa ratio; FFR; Collateral circulation
MeSH Terms: conditions — Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a consensus diagnosis of chronic mesenteric ischemia: Patients with a consensus diagnosis of chronic mesenteric ischemia who are scheduled for endovascular treatment

SUMMARY:
Chronic mesenteric ischemia (CMI) is an incapacitating disease with a vast impact on quality of life due to severe abdominal pain after a meal, resulting in fear of eating and subsequent weight loss. CMI is most frequently caused by an atherosclerotic mesenteric artery stenosis, which is a frequent finding in the general population (6-29%). CMI is less prevalent due to an extensive collateral circulation protecting the gut against ischemia.

Hence, imaging alone cannot be relied upon, making the diagnosis of CMI challenging. Treatment decisions for atherosclerotic CMI are currently based on history, stenosis severity on imaging, and signs of mesenteric ischemia during a functional test. Yet, sufficiency of the collateral circulation cannot be assessed, resulting in substantial failure to recover from symptoms after stentplacement (27-31% in single vessel disease), unnecessary complications, and avoidable healthcare expenses. A retrospective cohort study by van Dijk et al. reports that intra-arterial pressure measurements could predict clinical success of mesenteric artery revascularization with an 86% sensitivity and 83% specificity, indicating that mesenteric artery pressure measurements could be a highly desired and promising tool for the assessment of hemodynamic and clinical relevance of a mesenteric artery stenosis. Which is sensible, since pressure gradients will only occur when both a severe mesenteric artery stenosis and an insufficient collateral circulation are present. Another advantages of pressure measurements is the ability to simulate the postprandial physiology, using nitroglycerin, enabling measurements when mesenteric blood flow is maximal. Intra-arterial pressure measurements are currently the most promising tool to guide clinical decision making in patients with suspected CMI and could result in major improvements in quality of life by improving clinical success of mesenteric artery revascularization, decreasing complication risks and decreasing healthcare costs by facilitating allocation of health care resources to those patients actually benefitting from treatment.

DETAILED DESCRIPTION:
Chronic mesenteric ischemia (CMI) is an incapacitating disease with a vast impact on quality of life due to severe abdominal pain after a meal, resulting in fear of eating and subsequent severe weight loss. CMI has an incidence of 9.2 per 100,000, which increases with age to up to 44.3 per 100,000 in persons of ≥80 years. These incidence rates are higher than the incidence rates of other more well-known diseases, such as esophageal cancer (4.3 per 100,000) or ruptured abdominal aortic aneurysms (7.0 per 100,000), and even approximates the incidence of Crohn's disease (10.9 per 100,000). The prevalence of atherosclerotic mesenteric artery stenosis, the leading cause of CMI, is even higher (6-29%). An extensive collateral circulation protects the gut against ischemia in the majority of patients. Hence, not all mesenteric artery stenoses result in CMI and only those stenoses that are hemodynamically significant should be treated. Treatment decisions for atherosclerotic CMI are currently based on history, stenosis severity on imaging, and signs of mesenteric ischemia during a functional test. However, sufficiency of the collateral circulation cannot be assessed, resulting in substantial failure of patient-reported symptom relief after stent placement (27-31% in single vessel disease), unnecessary complications and avoidable healthcare expenses.

The Dutch Mesenteric Ischemia Study group (DMIS) consists of experts in the field of CMI and aims to improve both the quality of care and the quality of life of CMI patients by initiating and designing studies to provide patient-centered and evidence-based solutions to pending challenges in the field of CMI. In recent years the DMIS has been searching for a reliable tool to assess hemodynamic significance of a mesenteric artery stenosis, while accounting for the collateral circulation, in order to guide treatment decisions and avoid clinically unbeneficial revascularization procedures. In a retrospective study flow velocities were increased in the unaffected mesenteric artery when either the CA or SMA were stenosed. The increased blood flow in the unaffected vessel could indicate a well-functioning collateral network where blood flow is rerouted to prevent chronic mesenteric ischemia.

Another retrospective cohort study reports that intra-arterial pressure measurements, using a 4Fr catheter, could predict clinical success of mesenteric artery revascularization with an 86% sensitivity and 83% specificity. In this retrospective study, pressure gradients were obtained after administration of a vasodilator. With these pressure measurements, the Pd/Pa ratio and the fractional flow reserve (FFR) were measured. The Pd/Pa ratio is the pressure distal to the stenosis divided by pressure in the aorta and the FFR is the Pd/Pa ratio under hyperemic conditions, after administration of a vasodilator. Mesenteric artery pressure measurements could be a promising tool for the assessment of hemodynamic and clinical relevance of mesenteric artery stenosis, since pressure gradients will only occur in mesenteric arteries with a severe stenosis and an insufficient collateral circulation.

The previously performed retrospective study yielded promising results, but had some methodological limitations. Pressure measurements in the conducted study were only obtained in a subset of CMI patients by the decision of the interventional radiologist, with pressure measurements in general only performed when the radiologist was in doubt about the significance of the stenosis. This could have potentially led to selection bias and makes reproducibility of this study difficult to the general population of CMI patients as a whole. In the proposed study, the investigator will perform pressure measurements in the general population of CMI patients with a consensus diagnosis of CMI who are scheduled for endovascular treatment, hypothesizing that stenosis grade (%) alone cannot predict hemodynamic significance accurately. By obtaining pressure measurements in all CMI patients, including borderline, high-grade stenoses and occlusions, the investigators aim to evaluate the (in)sufficiency of the mesenteric collateral network by measuring pressure gradients over the stenotic lesion. The investigators hope such pressure gradients can predict clinical treatment success for all CMI patients. If positive results are obtained in this study, the investigators hope these measurements can serve as a decision-making tool in suspected CMI patients (to stent or not to stent).

In an in-vitro study (currently under submission) in which postprandial states in the superior mesenteric artery (SMA) and celiac artery (CA) were simulated, pressure measurements were obtained using a 4Fr macrocatheter, microcatheter and pressure wire. It showed that especially for a stenosis ≥75% or a longer stenosis, the 4Fr catheter tended to overestimate the fractional flow reserve (FFR) when compared to the microcatheter, due to partial obstruction of the residual vessel lumen by the relatively large size of the 4Fr catheter compared to microcatheter or pressure wire. Taking this into consideration together with a wider applicability and lower costs, they recommended the microcatheter for clinical use.

In addition, intra-arterial stress pressure measurements with a vasodilator (nitroglycerin) could make the measurements more reliable, since intestinal ischemia mainly occurs after a meal when blood flow is maximal and expected to increase by 30-150%. Ischemia in CMI is thus temporary and this dynamic process causes false negative tests when blood flow is not maximal. Intra-arterial injection of nitroglycerin is able to increase the mesenteric blood flow, thereby challenging the compensatory capacity of the mesenteric circulation and predicting clinical success of revascularization. In a retrospective study, the Pd/Pa ratio after administration of nitroglycerin yielded the most promising results with the highest sensitivity and specificity.

Intra-arterial nitroglycerin is already routinely administered during coronary angiography for cardiology patients. Moreover, intra-arterial vasodilators can be used as treatment for acute nonocclusive mesenteric ischemia (NOMI). In the retrospective study, no adverse events related to intra-arterial nitroglycerin had occurred, making intra-arterial pressure measurements a safe and useful tool to guide future treatment decisions (to stent or not to stent). Successful implementation of this strategy could result in a substantial reduction of the number of unbeneficial mesenteric artery revascularizations, thereby avoiding potential loss of quality of life due to complications and a reduction of healthcare expenses.

Intra-arterial pressure measurements could also enlighten the debate on other topics regarding mesenteric artery revascularization. Current guidelines define a stenosis severity of ≥70% as significant in single vessel disease, while a ≥50% stenosis of the SMA is considered significant when accompanied by a ≥70% stenosis of the CA. These definitions are mainly based on expert opinion and cannot be supported with solid evidence. Intra-arterial pressure measurements could prove whether use of the current definitions should be continued or whether the definitions should be revised. The latter seems more probable, since hemodynamic significance of a mesenteric artery stenosis depends on a combination of both stenosis severity and the compensatory capacity of the collateral circulation, which cannot be assessed on computed tomography angiography (CTA) or magnetic resonance angiography (MRA). A future definition could state that pressure measurements are mandatory in all patients to confirm that revascularization is indicated.

The current recommendation to revascularize both mesenteric arteries in patients with multivessel disease of CA and SMA is another example of a recommendation that could be revised based on results of intra-arterial pressure measurements. Pressure measurements could identify those patients in whom stenting of both vessels is indicated. Measurement of normal pressures in the CA, after SMA revascularization, suggests that the CA stenosis is no longer hemodynamically relevant. Revascularization of the CA is in this case no longer indicated and both the possible complications of CA revascularization and the unneeded expenses of CA stenting can be avoided.

Intra-arterial pressure measurements are currently the most promising tool to guide clinical decision-making in patients with suspected CMI. Implementation of pressure measurements could result in major improvements in quality of life by tailoring treatment to the patient's needs, thereby improving the clinical success of mesenteric artery revascularization and decreasing complication risks. This will ultimately result in a reduction of population-based healthcare costs by facilitating allocation of healthcare resources to those patients actually benefitting from treatment. The DMIS has designed a multicenter study to determine the predictive value of intra-arterial pressure measurements after administration of nitroglycerin using a microcatheter to predict clinical success of mesenteric artery revascularization, to set an optimal cut-off for the guidance of treatment decisions, and to determine cost-effectiveness of future clinical implementation of intra-arterial pressure measurements.

Primary Objective:

- To assess the predictive performance of the Pd/Pa ratio after administration of a vasodilator to predict the clinical success of mesenteric artery stenting

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic mesenteric ischemia (CMI) and scheduled for endovascular procedure of the mesenteric arteries
* Age ≥18 years of age
* Patients who gave informed consent

Exclusion Criteria:

* Patients presenting with acute mesenteric ischemia
* Common origin of the SMA and CA (normal variant)
* Patients unable to give informed consent
* Pregnancy
* Other criteria the physician considers not compatible with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing an interventional or diagnostic endovascular procedure of the mesenteric arteries are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Pd/Pa ratio after administration of a vasodilator and its association with clinical success of mesenteric artery stenting | From enrollment to 3 months after treatment
  Pd/Pa ratio after administration of a vasodilator and its association with clinical success of mesenteric artery stenting

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Erasmus University Medical Centre Rotterdam, Rotterdam, South Holland
  - Franciscus, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Petersen AS, Kolkman JJ, Meerwaldt R, Huisman AB, van der Palen J, Zeebregts CJ, Geelkerken RH. Mesenteric stenosis, collaterals, and compensatory blood flow. J Vasc Surg. 2014 Jul;60(1):111-9, 119.e1-2. doi: 10.1016/j.jvs.2014.01.063. Epub 2014 Mar 18. PMID 24650741
- [Background] Sadiq I, Chamakura S, Siddiqi S, Margey R, Azemi T. Use of fractional flow reserve in the assessment of chronic mesenteric ischemia. Vasc Med. 2014 Jun;19(3):182-188. doi: 10.1177/1358863X14529617. Epub 2014 May 30. PMID 24879713
- [Background] Takiguchi T, Nakajima M, Ohbe H, Sasabuchi Y, Matsui H, Fushimi K, Kim S, Yokota H, Yasunaga H. Vasodilator Therapy and Mortality in Nonocclusive Mesenteric Ischemia: A Nationwide Observational Study. Crit Care Med. 2020 May;48(5):e356-e361. doi: 10.1097/CCM.0000000000004255. PMID 32044841
- [Background] Twiner MJ, Hennessy J, Wein R, Levy PD. Nitroglycerin Use in the Emergency Department: Current Perspectives. Open Access Emerg Med. 2022 Jul 9;14:327-333. doi: 10.2147/OAEM.S340513. eCollection 2022. PMID 35847764
- [Background] Boyer N, Beyer A, Gupta V, Dehghani H, Hindnavis V, Shunk K, Zimmet J, Yeghiazarians Y, Ports T, Boyle A. The effects of intra-arterial vasodilators on radial artery size and spasm: implications for contemporary use of trans-radial access for coronary angiography and percutaneous coronary intervention. Cardiovasc Revasc Med. 2013 Nov-Dec;14(6):321-4. doi: 10.1016/j.carrev.2013.08.009. Epub 2013 Oct 2. PMID 24095616
- [Background] Bertrand OF, Rao SV, Pancholy S, Jolly SS, Rodes-Cabau J, Larose E, Costerousse O, Hamon M, Mann T. Transradial approach for coronary angiography and interventions: results of the first international transradial practice survey. JACC Cardiovasc Interv. 2010 Oct;3(10):1022-31. doi: 10.1016/j.jcin.2010.07.013. PMID 20965460
- [Background] Pillai AK, Kalva SP, Hsu SL, Walker TG, Silberzweig JE, Annamalai G, Baerlocher MO, Mitchell JW, Midia M, Nikolic B, Dariushnia SR; Society of Interventional Radiology Standards of Practice Committee. Quality Improvement Guidelines for Mesenteric Angioplasty and Stent Placement for the Treatment of Chronic Mesenteric Ischemia. J Vasc Interv Radiol. 2018 May;29(5):642-647. doi: 10.1016/j.jvir.2017.11.024. Epub 2018 Mar 21. No abstract available. PMID 29574024
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Garcia LA, Carrozza JP Jr. Physiologic evaluation of translesion pressure gradients in peripheral arteries: comparison of pressure wire and catheter-derived measurements. J Interv Cardiol. 2007 Feb;20(1):63-5. doi: 10.1111/j.1540-8183.2007.00213.x. PMID 17300406
- [Background] Imbesi SG, Kerber CW. Pressure Measurements across Vascular Stenoses. Practice and Pitfalls. Interv Neuroradiol. 1999 Jun 30;5(2):139-44. doi: 10.1177/159101999900500205. Epub 2001 May 15. PMID 20670502
- [Background] Moneta GL, Yeager RA, Dalman R, Antonovic R, Hall LD, Porter JM. Duplex ultrasound criteria for diagnosis of splanchnic artery stenosis or occlusion. J Vasc Surg. 1991 Oct;14(4):511-8; discussion 518-20. PMID 1920649
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Bjorck M, Koelemay M, Acosta S, Bastos Goncalves F, Kolbel T, Kolkman JJ, Lees T, Lefevre JH, Menyhei G, Oderich G, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Sanddal Lindholt J, Vega de Ceniga M, Vermassen F, Verzini F, Document Reviewers, Geelkerken B, Gloviczki P, Huber T, Naylor R. Editor's Choice - Management of the Diseases of Mesenteric Arteries and Veins: Clinical Practice Guidelines of the European Society of Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2017 Apr;53(4):460-510. doi: 10.1016/j.ejvs.2017.01.010. No abstract available. PMID 28359440
- [Background] van Dijk LJD, Harki J, van Noord D, Verhagen HJM, Kolkman JJ, Geelkerken RH, Bruno MJ, Moelker A; Dutch Mesenteric Ischemia Study group (DMIS). Covered stents versus Bare-metal stents in chronic atherosclerotic Gastrointestinal Ischemia (CoBaGI): study protocol for a randomized controlled trial. Trials. 2019 Aug 20;20(1):519. doi: 10.1186/s13063-019-3609-8. PMID 31429792
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Brazier J, Roberts J, Deverill M. The estimation of a preference-based measure of health from the SF-36. J Health Econ. 2002 Mar;21(2):271-92. doi: 10.1016/s0167-6296(01)00130-8. PMID 11939242
- [Background] Mensink PB, Moons LM, Kuipers EJ. Chronic gastrointestinal ischaemia: shifting paradigms. Gut. 2011 May;60(5):722-37. doi: 10.1136/gut.2009.199695. Epub 2010 Nov 29. PMID 21115543
- [Background] van Dijk LJD, Terlouw LG, van Noord D, Bijdevaate DC, Bruno MJ, Moelker A. Endovascular Pressure Measurements to Assess the Functional Severity of Mesenteric Arterial Stenoses. J Vasc Interv Radiol. 2020 Mar;31(3):430-437. doi: 10.1016/j.jvir.2019.10.019. Epub 2020 Jan 29. PMID 32007405
- [Background] van Dijk LJ, van Noord D, de Vries AC, Kolkman JJ, Geelkerken RH, Verhagen HJ, Moelker A, Bruno MJ. Clinical management of chronic mesenteric ischemia. United European Gastroenterol J. 2019 Mar;7(2):179-188. doi: 10.1177/2050640618817698. Epub 2018 Dec 4. PMID 31080602
- [Background] van Petersen AS, Kolkman JJ, Gerrits DG, van der Palen J, Zeebregts CJ, Geelkerken RH; Dutch Mesenteric Ischemia Study Group. Clinical significance of mesenteric arterial collateral circulation in patients with celiac artery compression syndrome. J Vasc Surg. 2017 May;65(5):1366-1374. doi: 10.1016/j.jvs.2016.11.052. Epub 2017 Mar 2. PMID 28259570
- [Background] van den Heuvel TRA, Jeuring SFG, Zeegers MP, van Dongen DHE, Wolters A, Masclee AAM, Hameeteman WH, Romberg-Camps MJL, Oostenbrug LE, Pierik MJ, Jonkers DM. A 20-Year Temporal Change Analysis in Incidence, Presenting Phenotype and Mortality, in the Dutch IBDSL Cohort-Can Diagnostic Factors Explain the Increase in IBD Incidence? J Crohns Colitis. 2017 Oct 1;11(10):1169-1179. doi: 10.1093/ecco-jcc/jjx055. PMID 28430884
- [Background] Howard DP, Banerjee A, Fairhead JF, Handa A, Silver LE, Rothwell PM; Oxford Vascular Study. Age-specific incidence, risk factors and outcome of acute abdominal aortic aneurysms in a defined population. Br J Surg. 2015 Jul;102(8):907-15. doi: 10.1002/bjs.9838. Epub 2015 May 7. PMID 25955556
- [Background] Terlouw LG, Verbeten M, van Noord D, Brusse-Keizer M, Beumer RR, Geelkerken RH, Bruno MJ, Kolkman JJ; Dutch Mesenteric Ischemia Study Group. The Incidence of Chronic Mesenteric Ischemia in the Well-Defined Region of a Dutch Mesenteric Ischemia Expert Center. Clin Transl Gastroenterol. 2020 Aug;11(8):e00200. doi: 10.14309/ctg.0000000000000200. PMID 32955192
- [Background] Blauw JTM, Pastoors HAM, Brusse-Keizer M, Beuk RJ, Kolkman JJ, Geelkerken RH, For The Dutch Mesenteric Ischemia Study Group. The Impact of Revascularisation on Quality of Life in Chronic Mesenteric Ischemia. Can J Gastroenterol Hepatol. 2019 Nov 12;2019:7346013. doi: 10.1155/2019/7346013. eCollection 2019. PMID 31781520
- [Background] Alahdab F, Arwani R, Pasha AK, Razouki ZA, Prokop LJ, Huber TS, Murad MH. A systematic review and meta-analysis of endovascular versus open surgical revascularization for chronic mesenteric ischemia. J Vasc Surg. 2018 May;67(5):1598-1605. doi: 10.1016/j.jvs.2017.12.046. Epub 2018 Mar 20. PMID 29571626
- [Background] Terlouw LG, Moelker A, Abrahamsen J, Acosta S, Bakker OJ, Baumgartner I, Boyer L, Corcos O, van Dijk LJ, Duran M, Geelkerken RH, Illuminati G, Jackson RW, Karkkainen JM, Kolkman JJ, Lonn L, Mazzei MA, Nuzzo A, Pecoraro F, Raupach J, Verhagen HJ, Zech CJ, van Noord D, Bruno MJ. European guidelines on chronic mesenteric ischaemia - joint United European Gastroenterology, European Association for Gastroenterology, Endoscopy and Nutrition, European Society of Gastrointestinal and Abdominal Radiology, Netherlands Association of Hepatogastroenterologists, Hellenic Society of Gastroenterology, Cardiovascular and Interventional Radiological Society of Europe, and Dutch Mesenteric Ischemia Study group clinical guidelines on the diagnosis and treatment of patients with chronic mesenteric ischaemia. United European Gastroenterol J. 2020 May;8(4):371-395. doi: 10.1177/2050640620916681. Epub 2020 Apr 16. PMID 32297566